CLINICAL TRIAL: NCT01481272
Title: A Phase II Trial on Ofatumumab With IVAC Salvage Chemotherapy in Diffuse Large B Cell Lymphoma Patients Progressing or Relapsed After Prior R-CHOP Treatment Not Suitable for Autologous Stem Cell Transplant
Brief Title: Ofatumumab With IVAC Salvage Chemotherapy in Diffuse Large B Cell Lymphoma Patients
Acronym: PLRG8
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polish Lymphoma Research Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLRG8 (OMB114361); 2010-023568-42 (EudraCT Number)
Record Dates: First submitted 2011-11-14; First posted 2011-11-29 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Salvage therapy in DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ofatumumab; Etoposide; Ifosfamide; Mesna; Cytarabine; Methotrexate; Leucovorin; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- O-IVAC (Experimental): Ofatumumab Etoposide Ifosfamide Mesna Cytarabine Methotrexate Leukovorin Granulocyte-Colony Stimulating Factor
  Interventions: Drug: Ofatumumab; Drug: Etoposide; Drug: Ifosfamid; Drug: Mesna; Drug: Cytarabine; Drug: Methotrexate; Drug: Leukovorin; Drug: Granulocyte-Colony Stimulating Factor

INTERVENTIONS:
Drug: Ofatumumab — 1000 IV, according to detailed instruction included in the protocol, on day 1 of each 21-day cycle, maximum 6 cycles
  Other Names: Arzerra
Drug: Etoposide — 60mg/m2 IV, daily over 1 hour, on days 1-5 of 21-day cycle, maximum 6 cycles
  Other Names: VePesid
Drug: Ifosfamid — 1500mg/m2 or 1000mg/m2 (patients >/=60 years), IV, daily over 1 hour, on 1-5 days of each 21-day cycle, maximum 6 cycles
  Other Names: Ifex
Drug: Mesna — 300mg/m2 or 200mg/m2 (patients >/=60 years), IV, over 1 hour, mixed with ifosfamid then 900mg/m2 or 600mg/m2 (patients >/=60 years)over 12 hour or by local practice, on 1-5 days of each 21 day cycle, maximum 6 cycles
  Other Names: Mesnex
Drug: Cytarabine — 2g/m2 or 0,5-1g/m2 (patients >/= 60 years), IV, over 3 hours, 12 hourly (total of 4 doses), on days 1-2 of each 21 day cycle, maximum 6 cycles
  Other Names: Cytosar
Drug: Methotrexate — 12mg, it, on day 5 of each 21 days cycle, maximum 6 cycles
  Other Names: Methotrexat Ebeve
Drug: Leukovorin — 15mg, po 24 hours after methotrexate it
  Other Names: Folinic Acid
Drug: Granulocyte-Colony Stimulating Factor — 5 microgram/kg or 263 microgram ampoule, sc, daily, starting on day 7 of each 21 day cycle, until ANC>1.0x109/l
  Other Names: Filgrastim

SUMMARY:
It is expected that addition of anti-CD20 antibody - ofatumumab would enhance the activity of the etoposide+ifosphamide with mesna+cytarabine+methotrexate+lenograstim or filgrastim (IVAC) regimen. This study is planned to determine the efficacy and safety of ofatumumab in combination with IVAC chemotherapy in patients with CD20 positive diffuse large B cell lymphoma progressing or relapsed after prior R-CHOP chemotherapy not suitable for Autologous Stem Cell Transplant (ASCT).

DETAILED DESCRIPTION:
The purpose of this study is to assess the Overall Response Rate (ORR) = Complete Response (CR) + Partial Response (PR) in adult Diffuse Large B Cell Lymphoma (DLBCL) patients progressing or relapsed after prior R-CHOP treatment not suitable for ASCT treated with O-IVAC salvage chemotherapy regimen. The secondary objective is the evaluation of progression-free survival (PFS), event-free survival (EFS), overall survival (OS), safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients under consideration for participation in this study must meet all of the following inclusion criteria:
* Histologically confirmed CD20 positive diffuse large B-cell lymphoma.
* Progressing or relapsed following prior treatment including but not limited to rituximab-CHOP chemotherapy regimen.
* Not suitable for ASCT (age > 60 years, PS ≥ 2, prior ASCT as a part of the previous treatment for DLBCL, and/or other medical conditions that unable the patients to undergo the ASCT, e.g. NYHA II, creatinine clearance < 50 mL/min).
* Age ≥ 18 years.
* ECOG/ WHO performance status grades 0 - 3.
* Resolution of toxicities from previous therapy to grade ≤ 1.
* Written signed and dated informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Known or suspected hypersensitivity to study treatments.
* Prior treatment with anti-CD20 monoclonal antibodies with the exception of rituximab.
* Screening laboratory values:

  * platelets < 75 x 109/L (unless due to DLBCL involvement of the bone marrow),
  * neutrophils < 1.5 x 109/L (unless due to DLBCL involvement of the bone marrow),
  * creatinine > 2.0 times upper normal limit (unless normal creatinine clearance),
  * total bilirubin >1.5 times upper normal limit (unless due to DLBCL involvement of liver or a known history of Gilbert's disease),
  * ALT > 2.5 times upper normal limit (unless due to DLBCL involvement of liver),
  * alkaline phosphatase > 2.5 times upper normal limit (unless due to DLBCL involvement of the liver or bone marrow).
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrolment, whichever is longer, or currently participating in any other interventional clinical study.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequel.
* Known HIV positive.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Positive serology for Hepatitis B (HB).
* Positive serology for hepatitis C (HC).
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy.
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-11; Primary Completion 2017-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 12 months post-therapy
  Complete response + partial response

SECONDARY OUTCOMES:
Progression-free survival | 12 month post-therapy
  Staying free of disease progression
Event-free survival | 12 month post-therapy
  Staying free of event such as disease progression, relapse, death, starting new anticancer therapy, patient's refusal to continue study treatment, Serious Adverse Event that causes discontinuation of study treatment
Overall survival | 12 months post-therapy
  Time since entering the study till death of any reason
Number of participants with adverse events as a measure of safety and tolerability | 12 months post-therapy
  Reporting Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jan Walewski, Prof., Study Chair — CENTRUM ONKOLOGII - INSTYTUT im. Marii Skłodowskiej-Curie ul. W.K. Roentgena 5, 02-781 Warszawa; Krzysztof Warzocha, Prof., Principal Investigator — Instytut Hematologii i Transfuzjologii, 02-776 Warszawa ul. Indiry Gandhi 14; Andrzej Hellmann, Prof., Principal Investigator — Klinika Hematologii i Tranplantologii, Uniwersyteckie Centrum Medyczne, ul. Dębinki 7, 80-952 Gdańsk; Andrzej Pluta, Prof., Principal Investigator — Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny im. ks. Bronisława Markiewicza, ul. ks. Bielawskiego 18, 36-200 Brzozów; Andrzej Lange, Prof., Principal Investigator — Dolnośląskie Centrum Transplantacji Komórkowych, 53-439 Wrocław, ul. Grabiszyńska105; Wanda Knopinska-Posluszny, MD PhD, Principal Investigator — Oddz. Hematologii, Samodzielny Publiczny ZOZ MSW z Warminsko-Mazurskim Centrum Onkologii w Olsztynie; ul.Wojska Polskiego 37, 10-228 Olsztyn; Sebastian Giebel, Prof., Principal Investigator — Klinika Transplantacji Szpiku i Onkohematologii, Centrum Onkologii Instytut im. M. Sklodowskiej-Curie w Gliwicach; al. Wybrzeże Armii Krajowej 15, 44-101 Gliwice; Jan M Zaucha, Prof., Principal Investigator — Oddz. Onkologii i Radioterapii, Szpital Morski im. PCK; ul. Powstania Styczniowego 1, 81-519 Gdynia
Locations (8):
- Poland (8):
  - Dolnośląskie Centrum Transplantacji Komórkowych, Wroclaw, Lower Silesian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Centrum Onkologii - Istytut im. M.Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onkologiczny im. ks. Bronisława Markiewicza, Brzozów, Podkarpackie Voivodeship
  - Uniwersyteckie Cenrum Medyczne, Gdansk, Pomeranian Voivodeship
  - Szpital Morski im. PCK Oddz. Onkologii i Radioterapii, Gdynia, Pomeranian Voivodeship
  - Klinika Transplantacji Szpiku i Onkohematologii; Centrum Onkologii Instytut im. M.Sklodowskiej-Curie, Oddz. w Gliwicach, Gliwice, Silesian Voivodeship
  - Oddz. Hematologii, Samodzielny Publiczny ZOZ MSW z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship

IPD SHARING:
Plan to Share IPD: No